CLINICAL TRIAL: NCT03077503
Title: Comparison of Dexmedetomidine and Fentanyl to Prevent Hemodynamic Response to Skull Pins Application in Neurosurgery:Double Blind Randomized Controlled Trial
Brief Title: Comparison of Dexmedetomidine and Fentanyl to Prevent Hemodynamic Response to Skull Pins Application
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Clinical Assistant Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HE581303
Record Dates: First submitted 2017-03-04; First posted 2017-03-13 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Hemodynamic Response; Skull Pins Application
Keywords: Hemodynamic response; Skull pins application; Dexmedetomidine; Fentanyl
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded controlled trial was conducted from September 2015 to September 2016 in Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Thailand. Sixty patients who underwent craniotomy with insertion of skull pin were randomly allocated into group A and B. After patients entered the operative room, blood pressure and heart rate were measured (T1) then repeated measurement again (T2) when started induction, intubation and infusion dexmedetomidine 1 µg/kg over 10 min infusion in group A whereas group B received normal saline. At 3 minutes before skull pin insertion (T3), patient in group B received a single bolus of fentanyl 1 µg/kg whereas group A received normal saline. Then hemodynamic responses were recorded and repeated again at one minute before skull pin insertion (T4). Blood pressure and heart rate were observed at the time of skull pin insertion (T5) then repeated every 1 minutes after skull pin application until 5 minutes (T6 - T10).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After written informed consents were obtained, all participant was blinded from the study drug. The study drugs (dexmedetomidine and fentanyl) were prepared by anesthetist nurse who not involved in the study. Dexmedetomidine was labeled with group A whereas fentanyl was labeled with group B. The study drug was administrated by the blinded anesthiologist. Blood pressure, mean arterial pressure, and heart rate were recorded by same blinded anesthesiologist
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Group A) (Experimental): In induction period, group A received dexmedetomidine 1 µg/kg diluted to 20 ml with 0.9% normal saline 10 minute through a syringe pump. Three minutes before application of skull pins, group A received infusion of 2 ml of 0.9% normal saline.
  Interventions: Drug: Dexmedetomidine; Drug: 0.9% normal saline; Device: Skull pins
- Fentanyl (group B) (Active Comparator): In induction period, group B received 20ml of 0.9% normal saline.Three minutes before application of skull pins, group B received infusion of fentanyl 1 µg/kg diluted to 2 ml with 0.9% normal saline
  Interventions: Drug: Fentanyl; Drug: 0.9% normal saline; Device: Skull pins

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 1 µg/kg diluted to 20 ml with 0.9% normal saline was administration. If adverse events were occurred, the patient will receive rescue drugs.
  Other Names: precedex
  Arms: Dexmedetomidine (Group A)
Drug: Fentanyl — Fentanyl 1 µg/kg diluted to 2 ml with 0.9% normal saline was administration. If adverse events were occurred, the patient will receive rescue drugs.
  Arms: Fentanyl (group B)
Drug: 0.9% normal saline — 0.9% normal saline was use to dilute the study drugs
Device: Skull pins — Skull pins were use to stabilized the patent' s head during surgery
  Other Names: Mayfield

SUMMARY:
To compare the effect between dexmedetomidine and fentanyl for controlling the hemodynamic response to skull pins application

DETAILED DESCRIPTION:
A randomized, double-blinded controlled trial was conducted from September 2015 to September 2016 in Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Thailand. Sixty patients who underwent craniotomy with insertion of skull pin were randomly allocated into group A and B. After patients entered the operative room, blood pressure and heart rate were measured (T1) then repeated measurement again (T2) when started induction, intubation and infusion dexmedetomidine 1 µg/kg over 10 min infusion in group A whereas group B received normal saline. At 3 minutes before skull pin insertion (T3), patient in group B received a single bolus of fentanyl 1 µg/kg whereas group A received normal saline. Then hemodynamic responses were recorded and repeated again at one minute before skull pin insertion (T4). Blood pressure and heart rate were observed at the time of skull pin insertion (T5) then repeated every 1 minutes after skull pin application until 5 minutes (T6 - T10).

ELIGIBILITY:
Inclusion Criteria:

* patients who scheduled for elective craniotomy under general anesthesia
* patient with American Society of Anesthesiologists physical status classification of I and II

Exclusion Criteria:

* patients having body mass index more than 30 kg/m2, heart rate lower than 45 bpm, hypertension, ischemic heart disease, heart block, on beta adrenergic blockers, medication allergy including propofol, fentanyl, and dexmedetomidine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline in time frame before pin insertion (T1-T4) , time during pin insertion (T5), repeated measurement time every 1 minute until 5 minutes after pin applications (T6-T10).
  Blood pressure was recorded by the blinded anesthesiologist

SECONDARY OUTCOMES:
Change in mean arterial pressure | Baseline in time frame before pin insertion (T1-T4), time during pin insertion (T5), repeated measurement time every 1 minute until 5 minutes after pin applications (T6-T10).
  Mean arterial pressure was recorded by the blinded anesthesiologist
Change in heart rate | Baseline in time frame before pin insertion (T1-T4), time during pin insertion (T5), repeated measurement time every 1 minute until 5 minutes after pin applications (T6-T10).
  Heart rate was recorded by the blinded anesthesiologist
adverse events | Baseline in time frame before pin insertion (T1-T4), time during pin insertion (T5), repeated measurement time every 1 minute until 5 minutes after pin applications (T6-T10).
  Adverse events were recorded by the blinded anesthesiologist. Rescue drugs were give when adverse events were occurred. Rescue drug include propofol (for hypertension), ephedrine(for hypotension), esmolol (for tachycardia), atropine (for bradycardia)

CONTACTS AND LOCATIONS:
Overall Officials: Pornthep Kasemsiri, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

REFERENCES:
- [Result] Paul A, Krishna HM. Comparison between intravenous dexmedetomidine and local lignocaine infiltration to attenuate the haemodynamic response to skull pin head holder application during craniotomy. Indian J Anaesth. 2015 Dec;59(12):785-8. doi: 10.4103/0019-5049.171558. PMID 26903671